CLINICAL TRIAL: NCT01627639
Title: A Randomized Trial to Evaluate Effectiveness of Acetazolamide in COPD Patients Developing Metabolic Alkalosis During Invasive Mechanical Ventilation
Brief Title: Effectiveness of Acetazolamide for Reversal of Metabolic Alkalosis in Mechanically Ventilated Chronic Obstructive Pulmonary Disease Patients
Acronym: DIABOLO
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Ministry of Health, France (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AOM09109
Record Dates: First submitted 2012-04-02; First posted 2012-06-26 (Estimated); Last update posted 2015-10-06 (Estimated); Status verified 2015-10

CONDITIONS: Decompensated Chronic Obstructive Pulmonary Disease
MeSH Terms: interventions — Acetazolamide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Acetazolamide (Active Comparator): Acetazolamide (1 g IV per day or 2 g IV per day if coprescription of loop diuretics) or Placebo (saline serum) when pure or mixed metabolic alkalosis being present until planned extubation
  Interventions: Drug: Acetazolamide
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Acetazolamide — Acetazolamide (1 g IV per day or 2 g IV per day if coprescription of loop diuretics) or Placebo (saline serum) when pure or mixed metabolic alkalosis being present until planned extubation
  Arms: Acetazolamide
Drug: Placebo — Placebo
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine whether acetazolamide are effective to reduce the length of mechanical ventilation in decompensated Chronic Obstructive Pulmonary Disease (COPD) patients developing pure or mixed metabolic alkalosis.

DETAILED DESCRIPTION:
The purpose of this study is to determine whether acetazolamide is effective to reduce the length of mechanical ventilation in decompensated COPD patients developing pure or mixed metabolic alkalosis.

ELIGIBILITY:
Inclusion Criteria:

* Decompensated COPD on invasive mechanical ventilation Less than 24 hours

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 380 (Actual)
Dates: Start 2011-10; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
length of invasive mechanical ventilation | within the first 28 days after intubation

SECONDARY OUTCOMES:
Length of weaning from mechanical ventilation | once at the extubation or at day 28
  data retrieved once, at the extubation or at the end of invasive ventilation in the tracheotomy
weaning success | once at the end of ICU stay or at Day 28
  Data collected once at the end of ICU stay or at Day 28
numbers of nosocomial infections | every day during 28 days
  data retrieved every day, until extubation or at the end of invasive ventilation in the tracheotomy
length of ICU stay | once at the end of ICU stay or at Day 28
  Data collected once at the end of ICU stay or at Day 28
ICU mortality | once at the end of ICU stay or at Day 28
  Data collected once at the end of ICU stay or at Day 28

CONTACTS AND LOCATIONS:
Overall Officials: Christophe Faisy, MD, PhD, Principal Investigator — Medical Intensive Care Unit, European Georges Pompidou Hospital, Asssistance Publique - Hôpitaux de Paris, Paris Descartes University, Paris, FRance
Locations (1):
- Clinical Research Unit, European Georges Pompidou Hospital, Assistance Publique - Hôpitaux de Paris, Paris, France

REFERENCES:
- [Background] Heming N, Faisy C, Urien S. Population pharmacodynamic model of bicarbonate response to acetazolamide in mechanically ventilated chronic obstructive pulmonary disease patients. Crit Care. 2011;15(5):R213. doi: 10.1186/cc10448. Epub 2011 Sep 14. PMID 21917139
- [Background] Chang WT, Thayer DW. The cellulase system of a Cytophaga species. Can J Microbiol. 1977 Sep;23(9):1285-92. doi: 10.1139/m77-192. PMID 20217
- [Derived] Faisy C, Meziani F, Planquette B, Clavel M, Gacouin A, Bornstain C, Schneider F, Duguet A, Gibot S, Lerolle N, Ricard JD, Sanchez O, Djibre M, Ricome JL, Rabbat A, Heming N, Urien S, Esvan M, Katsahian S; DIABOLO Investigators. Effect of Acetazolamide vs Placebo on Duration of Invasive Mechanical Ventilation Among Patients With Chronic Obstructive Pulmonary Disease: A Randomized Clinical Trial. JAMA. 2016 Feb 2;315(5):480-8. doi: 10.1001/jama.2016.0019. PMID 26836730